CLINICAL TRIAL: NCT00198601
Title: Determination of Gentamicin Dosing in Neonatal Patients for Use in the Uniject Pre-filled Syringe [A Three-site Study at: 1) Dhaka Shishu Hospital, Dhaka Bangladesh; 2) Christain Medical Center, Vellore, India; and 3) Aga Khan University Medical Center, Karachi, Pakistan]
Brief Title: Determination of Gentamicin Dosing in Neonatal Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H.22.02.08.30.B1
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2018-04-20 (Actual); Status verified 2005-09

CONDITIONS: Infection
Keywords: meningitis; neonatal deaths; gentamicin; Uniject; aminoglycoside
MeSH Terms: conditions — Infections; Meningitis; Perinatal Death | interventions — Gentamicins

INTERVENTIONS:
Drug: Gentamicin in Uniject Pre-filled syringe

SUMMARY:
The purpose of this study is to determine what dosage of gentamicin for use in one-time administration device (Uniject) is appropriate.

DETAILED DESCRIPTION:
This study aims to verify dosages of gentamicin for use in Uniject, chosen based on a consideration of gentamicin pharmacokinetics, safety, efficacy, target population body weight, cost, feasibility and acceptability.

ELIGIBILITY:
Inclusion Criteria:

* infants with culture proven sepsis
* infants 2000-2499 at birth
* infants > 2500 gm at birth
* infants < 2000 gm at birth
* in study site areas: Pakistan, Bangladesh and India

Exclusion Criteria:

* infants w/o culture proven sepsis

Ages: 1 Minute to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-08; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

PRIMARY OUTCOMES:
Patients 2.0-2.24 kg high peak>12.0: 2/6 patients
Low peak<4.0: none
High trough > 2.0: 1/6 patients

SECONDARY OUTCOMES:
Patients 2.5-3.0 kg
High peak>12.0: 2/14 patients
Low peak <4.0: none
High trough>2.0:2/14 patients

CONTACTS AND LOCATIONS:
Overall Officials: Gary Darmstadt, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (3):
- Dhaka Shishu Hospital, Dhaka, Bangladesh
- Neonatal Intensive Care Unit - Christian Vellore Medical, Vellore, India
- Aga Khan, Karachi, Pakistan